CLINICAL TRIAL: NCT00758446
Title: A Double-blind, Randomized, Placebo-controlled, Cross-over, Allergen Challenge Study to Evaluate the Efficacy, Safety and Tolerability of BLX-028914 in Subjects With Allergic Rhinitis
Brief Title: Efficacy and Safety Study of BLX-028914 in Subjects With Allergic Rhinitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dart NeuroScience, LLC (Industry)
Collaborators: Orexo AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: OX914-001
Record Dates: First submitted 2008-09-22; First posted 2008-09-25 (Estimated); Last update posted 2013-03-13 (Estimated); Status verified 2013-03

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental): BLX-028914 50 mg
  Interventions: Drug: BLX-028914
- B (Experimental): BLX-028914 15 mg
  Interventions: Drug: BLX-028914
- C (Placebo Comparator): Placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: BLX-028914 — 50 mg capsules, p.o, daily, 14 days
  Arms: A
Drug: BLX-028914 — 15 mg capsules, p.o, daily, 14 days
  Arms: B
Drug: placebo — capsules, p.o, daily, 14 days
  Arms: C

SUMMARY:
This is a phase II study in patients with seasonal allergic rhinitis (SAR) and will compare the effect versus placebo of two different oral doses of BLX-028914 in an allergen challenge model. BLX-028914, a selective phosphodiesterase-4 (PDE4) inhibitor with a promising safety profile,is currently under development for treatment of airway diseases by Orexo AB, Sweden.

The aim of this study is to compare the effect, safety and tolerability of 14 days treatment with BLX-0289014 in patients with SAR in an allergen challenge model versus placebo.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 50 years of age (inclusive), male or female
* Body Mass Index (BMI) between 18 and 28 kg/m2 (inclusive)
* History of pollen-induced seasonal allergic rhinitis but otherwise healthy
* Positive skin prick test for timothy and/or birch allergen
* Sufficient reaction to nasally administered allergen at screening
* Signed informed consent obtained

Exclusion Criteria:

* Expected symptoms of seasonal allergic rhinitis during the study period
* Asthma
* Nasal anatomical deviations, ongoing nasal symptoms, ongoing upper respiratory tract infection
* Anti-allergy immunotherapy in the previous two years
* Extensive use of nasal sprays
* Any medication except for contraceptives, during their last five half- lives prior to the first treatment period except for occasional OTC analgesics
* Ingestion of grapefruit or grapefruit juice or herbal remedies (e.g. St John's-wort) that may effect the enzyme CYP3A4
* Smoking within 3 months of first treatment period
* Clinically significant laboratory findings
* Pregnant or breast feeding woman or woman of childbearing potential not using adequate birth control
* Known hypersensitivity to any constituent of the study medication or placebo
* Participation in any other investigational study in the last three months
* Subject anticipated not being able to adhere to study plan according to investigator judgement

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2008-09; Primary Completion 2008-12 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Post allergen challenge; Total Nasal Symptom Score(TNSS) | 10 minutes after allergen challenge

CONTACTS AND LOCATIONS:
Overall Officials: Lennart Greiff, MD, PhD, Principal Investigator — Department of otorhinolaryngology
Locations (1):
- Department of otorhinolaryngology, Lund, Sweden